CLINICAL TRIAL: NCT00393315
Title: P E P C A D II, The Paclitaxel-Eluting PTCA-Balloon Catheter in Coronary Artery Disease to Treat In-Stent Restenoses: A Comparison to the Paclitaxel-Eluting Taxus™ Stent. A Pilot Study
Brief Title: P E P C A D II, The Paclitaxel-Eluting PTCA-Balloon Catheter in Coronary Artery Disease to Treat In-Stent Restenoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Bruno Scheller, University Hospital, Saarland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBM-VS-53; PEPCAD II/CRI/05/-02/c-c
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: In-Stent Restenosis
Keywords: in stent restenosis; paclitaxel coated balloon catheter; pepcad; drug eluting balloon

INTERVENTIONS:
Device: paclitaxel coated balloon catheter

SUMMARY:
The aim of the study is to assess the safety and efficacy of the Paclitaxel-eluting PTCA-balloon in the treatment of in-stent restenoses in native coronary arteries with reference diameters between 2.5 mm and 3.5 mm and ≤ 22 mm in length for procedural success and preservation of vessel patency in comparison to the Paclitaxel-eluting Taxus™ stent.

DETAILED DESCRIPTION:
Background information:

Stent deployment for the treatment of coronary artery stenoses has evolved as the standard treatment in nearly all types of coronary lesions over the past two decades.The initial recurrence rate of bare stents in the range of 20 30 % in low risk stenoses has been further reduced by devices with passive coatings such as silicon carbide, heparin, phosphorylcholine, and carbon. The significant decline of in-stent restenoses (= ISR) to the order of 12 % was achieved by active coatings like the cell-cycle inhibitor sirolimus and to about 13.7 % by the cytotoxic paclitaxel. Taken into account the more than one million annual stent procedures performed worldwide even low recurrence rates will leave some hundred thousand repeat procedures annually. In the treatment of in-stent restenoses, however, approaches such as stand alone angioplasty with conventional balloons, the repeat use of bare stents, cutting balloon angioplasty, rotablation, and atherectomy have revealed unsatisfactory and often conflicting results. For brachytherapy the late loss was reported in the range from 0.22 +/- 0.84 mm to 0.73 +/- 0.79mm. Due to its disadvantages such as delayed endothelialization with ensuing late thrombosis cumulating in a 12-months cardiac event rate of up to 30% rising to 50% after five years, its decrease of benefit over time, and the cumbersome logistics at the sites and in the labs, brachytherapy is not considered as a valid approach of the future. Recently, the deployment of drug eluting stents into a restenotic device was associated with restenosis rates in the range from 4% to 30% suggesting some advantage over the aforementioned approaches. The wide range of the results and some late cardiac events still leave room for alternative methods such as the Paclitaxel-eluting PTCA balloon catheter.

Study Rationale The principle of the Paclitaxel-eluting PTCA balloon catheter is based on the antiproliferative mode of action of the compound, the latter being homogenously distributed along the entire length of the balloon and, hence, the vessel segment to be treated. This advantage is in particular relevant in comparison to drug eluting stents as are the lack of chronic mechanical alterations of the artery, the ease of access to the lesion, the obviation of adding another layer of metal to the lesion, and the presumably lower cost of the procedure. Data on the use of the Paclitaxel-eluting PTCA balloon catheter on the treatment of in-stent restenoses, however, are scant. In the animal model and according to unpublished results in humans, the proliferation induced by a Paclitaxel-eluting balloon catheter was significantly less compared to an uncoated balloon and to the Sirolimus-eluting Cypher™ stent.Therefore, it is prudent to compare the direct arterial application of Paclitaxel by means of the Paclitaxel-eluting PTCA balloon catheter versus the Paclitaxel-eluting Taxus™-stent as percutaneous transluminal treatment options of in-stent restenosis in human coronary arteries in a prospective randomized pilot study.

ELIGIBILITY:
Inclusion Criteria: Patient Related

* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Age at least 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6 months follow-up
* Patients must agree to undergo the 6 months angiographic follow-up and the 1 and 3 year clinical follow-up Inclusion Criteria: Lesion Related
* In-stent restenosis or Mehran type III stenoses reaching ≤ 2 mm into the adjacent native vessel of a metal stent (including passive coatings, exclusive of active coatings), i.e., no recurrence in the native vessel adjacent to the stent, after stent deployment in a native coronary artery (reference vessel between 2.5 and 3.5 mm, lesion length ≤ 22 mm as angiographically documented)
* Diameter stenosis pre procedure must be either at least 70 % or 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, scintigraphy, MRT, or suspected based on angina pectoris
* In the stent group, the target lesion must be treated with a single stent only (multiple stenting shifts the patient to the intention-to-treat group) Exclusion Criteria: Patient Related
* Patients with acute (< 24 h) or recent (48 hours) myocardial infarction, unstable angina pectoris (Braunwald class 3)
* Clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mmHg requiring inotropic support, IABP and/or fluid challenge)
* Patients with another coronary stent implanted previously into the target vessel
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min) and is therefore not eligible for angiography. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g., malignoma)
* Patients with any type of surgery during the week preceding the interventional procedure.
* Therapy with anticogulants Exclusion Criteria: Lesion Related
* Evidence of extensive thrombosis within target vessel before the intervention
* Side branch > 2 mm in diameter originating from the stent
* Bifurcate lesion
* Left main coronary artery stenosis
* Multilesion percutaneous coronary intervention within the same artery
* Percutaneous coronary intervention of venous graft
* Coronary artery occlusions of any type
* In-stent restenosis of a drug eluting stent (DES)
* In-segment stenosis of the native vessel within the 5 mm adjacent to the stent
* Lesion within 1 mm of vessel origin
* Exclusion Criteria Related to Concomitant Medication
* Patient is intolerant to aspirin and/or the ADP-antagonists clopidogrel or has a history of neutropenia, thrombocytopenia induced by ADP-antagonists, or severe hepatic dysfunction prohibiting the use of clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Late lumen loss at 6 months

SECONDARY OUTCOMES:
Procedural success
Occurrence of acute (up to 48 hours), subacute (up to 30 days), and late thrombosis
30-day MACE rate
Percent in-stent stenosis at 6 months
Percent in-segment stenosis at 6 months
In-stent late loss index at 6 months
Angiographic binary in-stent stenosis rate at 6 months
In-segment late loss index at 6 months
Angiographic binary in-segment stenosis rate at 6 months
Acute and cumulative MACE rate at 6 months
Cumulative MACE rate after one year
Cumulative MACE rate after three years
Indication for premature follow-up
Type of recurrence (Mehran-Classification)
Target vessel failure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Unverdorben, MD, PhD, Principal Investigator — Clinical Research Institute, Center for Cardiovascular Diseases, Heinz-Meise-Strasse 100, D-36199 Rotenburg a.d. Fulda, Germany
Locations (10):
- Germany (10):
  - Kerckhoff-Clinic Bad Nauheim, Bad Nauheim
  - Unfallkrankenhaus Berlin, Berlin
  - Medizinische Klinik, Kardiologie, Charité - Hochschulmedizin Berlin, Berlin
  - Klinikum Darmstadt, Medizinische Klinik I, Darmstadt
  - Medizinische Klinik, Kardiologie, St.-Johannes -Hospital, Dortmund
  - Städtische Kliniken Esslingen, Klinik für Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar
  - University of Saarland, Internal Medicine III, Homburg/Saar
  - I. Med. Abteilung, Krankenhaus Bogenhausen, München
  - University of Regensburg, Regensburg
  - Center for Cardiovascular Diseases, Cardiologic Clinic, Rotenburg A.d. Fulda

REFERENCES:
- [Background] Speck U, Scheller B, Abramjuk C, Breitwieser C, Dobberstein J, Boehm M, Hamm B. Neointima inhibition: comparison of effectiveness of non-stent-based local drug delivery and a drug-eluting stent in porcine coronary arteries. Radiology. 2006 Aug;240(2):411-8. doi: 10.1148/radiol.2402051248. PMID 16864669
- [Background] Custodis F, Scheller B, Laufs U. [Stable coronary artery disease -- case report]. Dtsch Med Wochenschr. 2006 Mar 17;131(11):554-5; quiz 563-4. doi: 10.1055/s-2006-933695. No abstract available. German. PMID 16538559
- [Background] Speck U, Scheller B, Abramjuk C, Bernhardt U. Drug delivery by angiographic contrast media: inhibition of restenosis. Acad Radiol. 2005 May;12 Suppl 1:S14-7. doi: 10.1016/j.acra.2005.02.017. No abstract available. PMID 16106539
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Speck U, Scheller B, Abramjuk C, Grossmann S, Mahnkopf D, Simon O. Inhibition of restenosis in stented porcine coronary arteries: uptake of Paclitaxel from angiographic contrast media. Invest Radiol. 2004 Mar;39(3):182-6. doi: 10.1097/01.rli.0000116125.96544.64. PMID 15076010
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Scheller B, Speck U, Romeike B, Schmitt A, Sovak M, Bohm M, Stoll HP. Contrast media as carriers for local drug delivery. Successful inhibition of neointimal proliferation in the porcine coronary stent model. Eur Heart J. 2003 Aug;24(15):1462-7. doi: 10.1016/s0195-668x(03)00317-8. PMID 12909076
- [Derived] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis: the three-year results of the PEPCAD II ISR study. EuroIntervention. 2015 Dec;11(8):926-34. doi: 10.4244/EIJY14M08_12. PMID 25169589
- [Derived] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593